CLINICAL TRIAL: NCT00717665
Title: Self-monitoring of Blood Pressure in Primary Care in Older Diabetic Patients With Uncontrolled Systolic Hypertension
Brief Title: Self-monitoring of Blood Pressure in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Dr. Alexander Logan, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESA 5970
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: High Blood Pressure
Keywords: Hypertension; Telemanagement; Home blood pressure monitoring; Self care
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, 1, I (Experimental)
  Interventions: Device: Home blood pressure tele-management system.
- A, 2, I (Active Comparator)
  Interventions: Other: Usual care.

INTERVENTIONS:
Device: Home blood pressure tele-management system. — Scheduled blood pressure monitoring with transmission of information to a central server for processing and disbursement.
  Arms: A, 1, I
Other: Usual care. — Patient self-monitoring of blood pressure with results taken by patient to the doctor at scheduled visits.
  Arms: A, 2, I

SUMMARY:
This study is an open randomized controlled trial of 12-month duration, which compares the use of a home blood pressure (BP) tele-management system to the usual approach of home BP monitoring in older diabetic patients with uncontrolled systolic hypertension. The purpose of this study is to determine whether home blood pressure tele-management system will markedly improve blood pressure control in a primary care setting.

DETAILED DESCRIPTION:
Hypertension is a major risk factor for renal and cardiovascular disease (CVD). While the health benefits of lowering blood pressure (BP) are well documented, population surveys have consistently found that less than a quarter of hypertensive patients have their BP under good control. Self-monitoring of BP at home has been extensively evaluated as a potentially useful tool to improve BP control and medication adherence in hypertensive patients.

We developed a user-centric home BP tele-management system. The system captures all home self-measured BP readings and requires patients to set jointly with their physician their BP treatment goal, home BP monitoring schedule and BP alert levels. The system tracks the frequency, date and time of home readings, generates messages for patients and reports for physicians indicating whether the BP treatment goal has been reached, and sends BP alerts and adherence reminders for BP readings to patients and clinical BP alerts and reports to physicians. Using an open, randomized controlled parallel group trial design, older diabetic patients with uncontrolled systolic hypertension, recruited from the practice of primary care physicians, will receive either usual care approach to home BP monitoring or care that incorporates the use of the home BP tele-management system. The primary outcome measure is the change in mean daytime systolic BP from baseline to the last (12-month) visit on 24-hour ambulatory. The secondary objective is to examine the psychosocial factors that may make it difficult for some patients to monitor their blood pressure at home. The rationale for including a psychological component in the study is that a critical component of the system is adherence to self-monitoring. While adherence can be automatically determined through the telemanagement system, the determinants of adherence to this behaviour have not been adequately assessed in the literature. To gain insights into this aspect of health behaviour we will measure psychological predictors using quantitative and qualitative techniques. Moreover, monitoring adherence with home BP monitoring will provide a proxy measure of acceptance of the system as a poor adherence rate would suggest that patients perceive it as a futile exercise, not leading to any changes in their care.

This study tests a novel approach to treat hypertension, a major health problem in diabetic patients. The information from this study will be invaluable for future health care planning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus (the onset of diabetes must have occurred on or after the age of 30 years and there is no history of diabetic ketoacidosis)
* Uncontrolled systolic hypertension (defined as a daytime systolic BP of 130 mm Hg or higher on 24-hour ambulatory)

Exclusion Criteria:

* Conditions making the patient unsuitable for study such as severe cognitive impairment, language difficulties (unable to speak and understand instructions in English), frequent (more than once per month for more than week) or prolonged (more than 2 months) trips away from home, homelessness, self-identified substance abuse, being pregnant, or unable to use home BP device;
* Life expectancy less than one year
* Coexisting conditions that require frequent (more than once a month) office visits or repeated (more than once in the past year) hospitalizations
* Atrial fibrillation or other cardiac arrhythmias requiring drug treatment
* Moderately severe chronic renal failure defined as estimated GFR less than 25 mL/min
* Myocardial infarction, episode of heart failure requiring hospitalization, or paralyzing stroke in the past year
* Having unstable angina
* Severe valvular heart diseases such as severe aortic stenosis
* Symptomatic orthostatic hypotension
* Refusal to sign consent form or to carry out the demands made by the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The change in mean daytime systolic BP from baseline to the last (12-month) visit on 24-hour ambulatory. | 1 year

SECONDARY OUTCOMES:
mean change in systolic and diastolic BP on 24-hour ambulatory and one-week home BP monitoring | from the baseline to the last (12-month) visit
mean change in daytime diastolic BP on 24-hour ambulatory BP monitoring | from the baseline to the last (12-month) visit
mean change in systolic and diastolic BP during the sleep period on 24-hour ambulatory BP monitoring | from the baseline to the last (12-month) visit
the proportion of patients at systolic BP goal, defined as <130 mmHg and diastolic BP goal, defined as <80 mm Hg, based on the 24-hour ambulatory BP and one-week home BP monitoring recording | one year
number and doses of different classes of antihypertensive medications | one year
average adherence rate with home BP monitoring | one year
the number of adherence reminders in the tele-management group over the course of the study | one year
the number of office visits of patients | during the one year study period
determinants of adherence to tele-monitoring | one year

CONTACTS AND LOCATIONS:
Overall Officials: Alexander G. Logan, MD, FRCP(C), Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Turnbull F; Blood Pressure Lowering Treatment Trialists' Collaboration. Effects of different blood-pressure-lowering regimens on major cardiovascular events: results of prospectively-designed overviews of randomised trials. Lancet. 2003 Nov 8;362(9395):1527-35. doi: 10.1016/s0140-6736(03)14739-3. PMID 14615107
- [Background] Wolf-Maier K, Cooper RS, Kramer H, Banegas JR, Giampaoli S, Joffres MR, Poulter N, Primatesta P, Stegmayr B, Thamm M. Hypertension treatment and control in five European countries, Canada, and the United States. Hypertension. 2004 Jan;43(1):10-7. doi: 10.1161/01.HYP.0000103630.72812.10. Epub 2003 Nov 24. PMID 14638619
- [Background] Logan AG, McIsaac WJ, Tisler A, Irvine MJ, Saunders A, Dunai A, Rizo CA, Feig DS, Hamill M, Trudel M, Cafazzo JA. Mobile phone-based remote patient monitoring system for management of hypertension in diabetic patients. Am J Hypertens. 2007 Sep;20(9):942-8. doi: 10.1016/j.amjhyper.2007.03.020. PMID 17765133
- [Derived] Logan AG, Irvine MJ, McIsaac WJ, Tisler A, Rossos PG, Easty A, Feig DS, Cafazzo JA. Effect of home blood pressure telemonitoring with self-care support on uncontrolled systolic hypertension in diabetics. Hypertension. 2012 Jul;60(1):51-7. doi: 10.1161/HYPERTENSIONAHA.111.188409. Epub 2012 May 21. PMID 22615116